CLINICAL TRIAL: NCT03711812
Title: SABRE: Serratus Anterior Block and Catheter Use in Rib Fractures in the Emergency Department
Brief Title: Serratus Anterior Block and Catheter Use in Rib Fractures in the Emergency Department
Acronym: SABRE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 232220
Record Dates: First submitted 2018-10-08; First posted 2018-10-18 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Anesthesia; Rib Fractures
Keywords: regional anaesthesia; rib fractures
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Anterior Plane Catheter (Active Comparator)
  Interventions: Procedure: Serratus Anterior Plane Catheter
- Thoracic Epidural (Placebo Comparator)
  Interventions: Procedure: Thoracic Epidural Catheter

INTERVENTIONS:
Procedure: Serratus Anterior Plane Catheter — Insertion of a Serratus Anterior Plane Catheter to establish a continuous analgesic block with a local anaesthetic infusion
  Arms: Serratus Anterior Plane Catheter
Procedure: Thoracic Epidural Catheter — Insertion of a Thoracic Epidural Catheter to establish a continuous analgesic block with a local anaesthetic infusion
  Arms: Thoracic Epidural

SUMMARY:
The main aim of this study is to determine whether Serratus Anterior Plane (SAP) blockade provides improved pain relief after rib fractures compared to epidural administration of local anaesthetic. The investigators aim to show that SAP catheters (SAPC) can be placed in more situations and are less operator-dependent then thoracic epidural anaesthesia (TEA). This reduces the waiting time required to achieve satisfactory analgesia in the patient. Optimal analgesia allows early respiratory physiotherapy and reduction in the complications of multiple rib fractures.

Pain from rib fractures is severe. The sensory nerves of the thoracic wall lie in the SAP and a single ultrasound-guided injection of local anaesthetic spreads widely and provides useful post-injury analgesia for several hours. If a catheter is left in the SAP, the nerve blockade can be maintained for several days.

Rib Fracture pain is traditionally treated with oral/ intravenous analgesics or TEA. Opiate analgesia via patient controlled analgesia (PCA) can work very well but it is associated with excessive sedation, constipation, nausea and vomiting. Continuous TEA is generally regarded as the gold standard but it demands monitoring by adequately trained ward staff and is commonly associated with high failure rates and increased risk of complications. SAPC has also been used when TEA and PCA were not desirable.

The primary outcome will be the amount of morphine analgesia required by the patient. Secondary outcomes will be pain scores (at rest and on movement), the side effects of morphine, complications of TEA/ SAPC, respiratory function changes and a quality of recovery assessment.

The control group will have an epidural block and catheter placed. The treatment group will have SAP blocks and catheters placed under ultrasound guidance. Both blocks will be tested to ensure good pain relief. To avoid potential confounding effects, oral painkillers will adhere strictly to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years suffering 2 or more rib fractures

Exclusion Criteria:

1. Significant renal dysfunction (baseline creatinine >150μmol/l - morphine contra- indicated)
2. Pregnancy
3. Patients with chronic pain on regular analgesic medication
4. Patients with significant coagulation abnormality (unsafe to site blocks)
5. Participation in another interventional study that will interact with this trial.
6. Patients unable to give informed consent
7. Hypersensitivity to local anaesthetic (or any other study drug).
8. Contraindication to NSAID (peptic ulceration or sensitive asthma)
9. Weight <50kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
intravenous morphine use via a patient controlled pump | 72 hours
  This will be measured as the total amount (in milligrams) of intravenous morphine used via a patient controlled pump in 72 hours.

SECONDARY OUTCOMES:
static and dynamic pain scores measurements | 72 hours
  This will be measured using a visual analogue scale from 0(no pain) to 10(unbearable pain). The measurement will be done whilst the patient is at rest and again on movement.
side effects/ complications of interventions | 72 hours
  The side effects and complications of either a thoracic epidural or serratus anterior plane block will be recorded. This includes failure to establish the block and/or catheter, decreased blood pressure, neurological sequelae, nausea and vomiting and itching.
spirometry | 72 hours
  Spirometry will be undertaken at the bedside and the tidal volumes will be recorded 3 times and the average taken of the 3 measurements.
quality of recovery assessment | 72 hours
  The quality of recovery (QoR) will be assessed using the QoR40. The QoR-40 is a 40-item questionnaire that provides a global score and subscores across five dimensions: patient support, comfort, emotions, physical independence, and pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom